CLINICAL TRIAL: NCT05098054
Title: Phase 1 Pharmacokinetics and Safety Study of Oral Soticlestat in Participants With Moderate or Mild Hepatic Impairment and Normal Hepatic Function
Brief Title: A Study of Soticlestat in Adults With Liver Failure Compared to Those With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-935-1010; 2021-006373-29 (EudraCT Number)
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — soticlestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1, Moderate HI: Soticlestat 300 mg (Experimental): Soticlestat 300 mg, tablets, orally, once on Day 1 to participant with moderate HI.
  Interventions: Drug: Soticlestat
- Arm 2, Mild HI: Soticlestat 300 mg (Experimental): Soticlestat 300 mg, tablets, orally, once on Day 1 to participant with mild HI.
  Interventions: Drug: Soticlestat
- Arm 3, Normal hepatic function: Soticlestat 300 mg (Experimental): Soticlestat 300 mg, tablets, orally, once on Day 1 to healthy participants.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablets.
  Other Names: TAK-935

SUMMARY:
The main aim is to check the effect of a single dose of soticlestat in adults with moderate or mild liver failure compared to healthy adults with normal liver function.

Participants will check into the study clinic for 8 days. During the stay, one oral dose of soticlestat will be given and the participant will be monitored. The clinic staff will follow up with the participant about a week after discharge from the clinic.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). The study will assess the safety and tolerability of single oral dose of soticlestat in participants with moderate or mild Hepatic Impairment (HI) compared to healthy participants matched by age (mean ±10 years), sex (±2 per sex), and body mass index (BMI, mean ±10 percent [%]) with normal hepatic function.

The study will enroll approximately 40 participants. Participants will be assigned to following study arms:

* Arm 1, Moderate HI: Soticlestat 300 milligram (mg) (Child-Pugh Class B)
* Arm 2, Mild HI: Soticlestat 300 mg (Child-Pugh Class A)
* Arm 3, Normal hepatic function: Soticlestat 300 mg

All participants will receive single oral dose of study drug. The data will be collected and stored in electronic case report form (eCRF).

This multi-center trial will be conducted in the United States and Hungary. The overall duration of the study is approximately 42 days. Participants will be followed up for 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria A. For Participants with Hepatic Impairment

1. Has a BMI greater than or equal to (>=) 18.0 and less than or equal to (<=) 40.0 kilogram per square meter (kg/m^2), at screening. At least 50% of the participants will be required to be of BMI >=18.0 and <=35.0 kg/m^2, at screening.

   * Supine blood pressure (BP) is >=80/40 millimeter of mercury (mmHg) (asymptomatic) and <=150/95 mmHg at screening;
   * Supine pulse rate (PR) is >=40 beats per minute (bpm) and <=99 bpm, at screening;
   * QT interval corrected for heart rate using Fridericia's formula (QTcF) is <=500 millisecond (msec) and ECG findings considered normal or not clinically significant by the Investigator or designee, at screening.
2. Must have had chronic HI for at least 3 months before screening, and the HI must be stable, that is, no significant changes in hepatic function in the 30 days preceding screening (or since the last visit if within 6 months before screening) and treatment with stable doses of medication. Has a score on the Child-Pugh Class at screening as follows:

   * (Arm 1) Moderate HI, Child-Pugh Class B: >=7 and <=9
   * (Arm 2) Mild HI, Child-Pugh Class A: >=5 and <=6
3. Should not have renal dysfunction as demonstrated by a relatively adequate renal function (creatinine clearance >=50 milliliter per minute [mL/min]), at screening.

B. For Healthy Participants

1. Has a BMI >=18.0 and <=40.0 kg/m^2, at screening. At least 50% of the participants will be required to be of BMI >=18.0 and <=35.0 kg/m^2, at screening. Healthy participants will be matched to hepatic impaired participants in this study by age (mean ±10 years), sex (±2 per sex), and BMI, mean ±10%.

   * Supine BP is >=90/40 mmHg and <=150/95 mmHg, at screening;
   * Supine PR is >=40 bpm and <=99 bpm, at screening;
   * QTcF is <=450 msec (males) or <=470 msec (females) and ECG findings considered normal or not clinically significant by the Investigator or designee, at screening;
   * Liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and total bilirubin <= the upper limit of normal (ULN) at screening and check-in.
2. Should not have renal dysfunction as demonstrated by a relatively adequate renal function (creatinine clearance >=60 mL/min), at screening.

C. For Participants with Hepatic Impairment and Healthy Participants

1. Continuous non-smoker or moderate smoker (<=10 cigarettes/day or the equivalent) before screening. Participant must agree to consume no more than 5 cigarettes or equivalent/day from the 7 days prior check-in and until discharge from the Clinical Research Unit (CRU).

Exclusion Criteria A. For Participants with Hepatic Impairment

1. Has history or presence of clinically significant medical or psychiatric condition or disease (aside from HI) or presence of psychotic disorders such as psychosis, delusions, or schizophrenia in the opinion of the Investigator or designee.
2. Has a history of liver or other solid organ transplant.
3. Positive result at screening for human immunodeficiency virus (HIV). Hepatitis B surface antigen (HBsAg) positive participants are allowed to be enrolled if Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is below 1000 copies per milliliter (/mL) in the plasma. Participants with moderate or mild HI who are positive for Hepatitis C virus antibodies (HCVAb) can be enrolled but must not have detectable Hepatitis C virus (HCV) ribonucleic acid (RNA) in the plasma.

B. For Healthy Participants

1. Has history or presence of clinically significant medical or psychiatric condition or disease or presence of psychotic disorders such as psychosis, delusions, or schizophrenia in the opinion of the Investigator or designee.
2. Positive results at screening for HIV, HBsAg, or HCV.

C. For Participants with Hepatic Impairment and Healthy Participants

1. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing.
2. Any positive responses on the Columbia-Suicide Severity Rating Scale (C-SSRS) or has a risk of suicide according to the Investigator's judgment based on the assessment of the C-SSRS at screening or check-in or has made a suicide attempt in the previous 12 months prior to dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- United States (5):
  - Velocity, Edgewater, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - GCP, St. Petersburg, Florida
  - Texas Liver Institute, San Antonio, Texas
- CRU Hungary Unit Pest Country Flor Ferenc Hospital, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6181de91eb0e19002afd69ee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 29 October 2021 to 07 June 2022.
Pre-assignment Details: Participants diagnosed with moderate/mild hepatic impairment (HI) compared to matched healthy participants with normal hepatic function received single dose of soticlestat. 1 with severe HI, 8 with moderate HI, 8 with mild HI and overall 19 participants with normal hepatic function (12 matched to moderate HI and 12 matched to mild HI participants) were enrolled. Five of same participants with normal hepatic function served as matched to moderate and mild HI.
Groups:
- Severe HI: Soticlestat 300 mg: Soticlestat 300 milligrams (mg), tablets, orally, once on Day 1 to participants with severe HI.
- Moderate HI: Soticlestat 300 mg: Soticlestat 300 mg, tablets, orally, once on Day 1 to participant with moderate HI.
- Mild HI: Soticlestat 300 mg: Soticlestat 300 mg, tablets, orally, once on Day 1 to participant with mild HI.
- Normal Hepatic Function: Soticlestat 300 mg: Soticlestat 300 mg, tablets, orally, once on Day 1 to healthy participants.
Period: Overall Study
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function: Soticlestat 300 mg
Started | 1 | 8 | 8 | 19
Completed | 1 | 8 | 8 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received the dose of soticlestat.
Groups:
- Severe HI: Soticlestat 300 mg: Soticlestat 300 mg, tablets, orally, once on Day 1 to participants with severe HI.
- Total: Total of all reporting groups
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function: Soticlestat 300 mg | Total
Number analyzed (Participants) | 1 | 8 | 8 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (NA) — Standard Deviation (SD) could not be calculated since only one participant was analyzed. | 59.4 (8.52) | 56.4 (10.03) | 58.2 (6.60) | 58.3 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 11 | 16
  Male | 1 | 5 | 6 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 5 | 11 | 23
  Not Hispanic or Latino | 0 | 2 | 3 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 5 | 6
  White | 1 | 7 | 7 | 14 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 8 | 8 | 19 | 36
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.460 (NA) — SD could not be calculated since one participant was analyzed. | 30.344 (4.0131) | 30.595 (4.9193) | 29.849 (1.7734) | 30.031 (3.1868)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 159.0 (NA) — SD could not be calculated since one participant was analyzed. | 166.1 (11.72) | 169.4 (13.39) | 167.5 (9.02) | 167.4 (10.41)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 66.90 (NA) — SD could not be calculated since one participant was analyzed. | 83.80 (14.289) | 88.51 (22.709) | 84.07 (11.124) | 84.52 (14.844)
Child-Pugh Score [Mean (Standard Deviation); unit: score on scale] — The Child-Pugh classification score was used to determine the severity of hepatic impairment. A participant was rated a score of 1 to 3 for each of the 5 categories: encephalopathy, ascites, bilirubin, albumin and INR. The total score was the sum of the scores for each category with a minimum of 5 and a maximum of 15. A participant would have a mild hepatic impairment with a Child-Pugh score of 5 to 6, a moderate impairment with a score of 7 to 9 and a severe impairment with a score of 10 to 15. A participant with normal hepatic function would have a score of 0 assigned. Population: Here 'number analyzed' signifies that participant who were evaluable for this baseline measure.
  score on scale
    number analyzed (Participants) | 1 | 8 | 8 | 0 | 17
    (all) | 10.00 (NA) — SD could not be calculated since one participant was analyzed. | 8.00 (0.926) | 5.50 (0.535) |  | 6.94 (1.64)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Soticlestat
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: Pharmacokinetic (PK) Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations) and were included in the statistical analyses. Five of the same participants with normal hepatic function served as matched to moderate and mild HI arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg: Soticlestat 300 mg, tablets, orally, once on Day 1 to healthy participants with normal hepatic function matched to moderate HI.
- Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg: Soticlestat 300 mg, tablets, orally, once on Day 1 to healthy participants with normal hepatic function matched to mild HI.
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg | Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg
Number analyzed (Participants) | 1 | 8 | 8 | 12 | 12
nanogram per milliliter (ng/mL) | 3230 (NA) — SD could not be calculated since only one participant was analyzed. | 3666 (130.9) | 1435 (109.9) | 1705 (81.9) | 986.9 (58.0)
Statistical Analysis 1: Comparison: Moderate HI: Soticlestat 300 mg vs Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg; Test type: Other; Geometric Least-squares mean(GLSM) Ratio = 214.93, 90% CI 2-sided [103.47 to 446.45] — Geometric least-squares means (LSMs) were calculated by exponentiating the LSMs from the mixed effects model. Geometric LSM Ratio (GMR) = 100*(Moderate HI/Normal Hepatic Function (Matched to Moderate HI)
Statistical Analysis 2: Comparison: Mild HI: Soticlestat 300 mg vs Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg; Test type: Other; GLSM Ratio = 145.42, 90% CI 2-sided [77.18 to 273.98] — Geometric LSMs were calculated by exponentiating the LSMs from the mixed effects model. Geometric LSM Ratio (GMR) = 100*(Mild HI/Normal Hepatic Function (Matched to Mild HI)

2. Primary Outcome: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Infinity for Soticlestat
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations) and were included in the statistical analyses. Five of the same participants with normal hepatic function served as matched to moderate and mild HI arms. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng•hr/mL)
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg | Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg
Number analyzed (Participants) | 1 | 8 | 6 | 10 | 11
nanogram*hour per milliliter (ng•hr/mL) | 2980 (NA) — SD could not be calculated since only one participant was analyzed. | 5760 (263.0) | 1539 (67.1) | 1925 (53.3) | 1182 (46.3)
Statistical Analysis 1: Comparison: Moderate HI: Soticlestat 300 mg vs Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg; Test type: Other; GLSM Ratio = 299.21, 90% CI 2-sided [111.75 to 801.17] — Geometric LSMs were calculated by exponentiating the LSMs from the mixed effects model. Geometric LSM Ratio (GMR) = 100*(Moderate HI/Normal Hepatic Function (Matched to Moderate HI)
Statistical Analysis 2: Comparison: Mild HI: Soticlestat 300 mg vs Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg; Test type: Other; GLSM Ratio = 130.25, 90% CI 2-sided [77.02 to 220.26] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for Soticlestat
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations) and were included in the statistical analyses. Five of the same participants with normal hepatic function served as matched to moderate and mild HI arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg | Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg
Number analyzed (Participants) | 1 | 8 | 8 | 12 | 12
ng*hr/mL | 2960 (NA) — SD could not be calculated since only one participant was analyzed. | 5732 (266.1) | 1522 (55.5) | 1812 (58.1) | 1126 (46.2)
Statistical Analysis 1: Comparison: Moderate HI: Soticlestat 300 mg vs Normal Hepatic Function (Matched to Moderate HI): Soticlestat 300 mg; Test type: Other; GLSM Ratio = 316.27, 90% CI 2-sided [117.68 to 849.97] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Mild HI: Soticlestat 300 mg vs Normal Hepatic Function (Matched to Mild HI): Soticlestat 300 mg; Test type: Other; GLSM Ratio = 135.26, 90% CI 2-sided [91.22 to 200.57] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE that started or worsened at the time of or after dosing of study drug.
Time Frame: From Day 1 up to 16 days after the last dose of study drug (up to Day 17)
Population: Safety analysis set included all participants who received the dose of soticlestat.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function: Soticlestat 300 mg
Number analyzed (Participants) | 1 | 8 | 8 | 19
Participants | 1 | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started from Day 1 up to 16 days after the last dose of study drug (up to Day 17)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Severe HI: Soticlestat 300 mg | Moderate HI: Soticlestat 300 mg | Mild HI: Soticlestat 300 mg | Normal Hepatic Function: Soticlestat 300 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/8 | 0/8 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/8 | 0/8 | 0/19
Other Adverse Events (participants affected / at risk) | 1/1 | 1/8 | 1/8 | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe HI: Soticlestat 300 mg (N=1) | Moderate HI: Soticlestat 300 mg (N=8) | Mild HI: Soticlestat 300 mg (N=8) | Normal Hepatic Function: Soticlestat 300 mg (N=19)
Alpha-1 acid glycoprotein increased (Investigations) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT05098054/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT05098054/SAP_001.pdf